CLINICAL TRIAL: NCT02495038
Title: Optimal Dose of Combination of Rocuronium and Cisatracurium: A Randomized Double-blinded Clinical Trial
Brief Title: Optimal Dose of Combination of Rocuronium and Cisatracurium
Acronym: CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Wooyoung Park, clinical assistant professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: combination P-1
Record Dates: First submitted 2015-06-04; First posted 2015-07-13 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-01

CONDITIONS: Chronic Otitis Media; Anesthesia
Keywords: combination; rocuronium; cisatracurium; neuromuscular blockade monitoring; drug synergism
MeSH Terms: interventions — cisatracurium; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intubating dose, Group I (No Intervention): combined ED95 rocuronium and ED95 cisatracurium
  ED95, dose causing on average 95% suppression of neuromuscular response.
- 10% reduction of combination of Esmeron® and Nimbex®, Group S (Experimental): This arm reduced 10% of combined ED95 rocuronium and ED95 cisatracurium
  Interventions: Drug: 10% reduction of combination of Esmeron® and Nimbex®
- 20% reduction of combination of Esmeron® and Nimbex®, Group L (Experimental): This arm reduced 20% of combined ED95 rocuronium and ED95 cisatracurium
  Interventions: Drug: 20% reduction of combination of Esmeron® and Nimbex®

INTERVENTIONS:
Drug: 10% reduction of combination of Esmeron® and Nimbex® — Patients were randomly assigned to each group by opening of sealed allocation envelope. After collection of data, allocation number was matched with each group. The participants matched at Group S were administered with NMBAs reduced 10% of each ED95. Before patients arrived in the operating room, rocuronium and cisatracurium were prepared by a nurse who was not involved in this study. Each drug dosage was determined by allocation number. The syringe containing each study drug was conveyed to the performer of this study as the status of shielding the scale. The syringes of rocuronium and cisatracurium used each other syringe.
  Other Names: Esmeron®, 74119419, ATC code:M03AC09; Nimbex®, 74500213, ATC code:M03AC11
  Arms: 10% reduction of combination of Esmeron® and Nimbex®, Group S
Drug: 20% reduction of combination of Esmeron® and Nimbex® — The participants matched at Group L were administered with NMBAs reduced 20% of each ED95.
  Other Names: Esmeron®, 74119419, ATC code:M03AC09; Nimbex®, 74500213, ATC code:M03AC11
  Arms: 20% reduction of combination of Esmeron® and Nimbex®, Group L

SUMMARY:
BACKGROUND: The combinations of rocuronium and cisatracurium have a synergic effect. The investigators studied whether the prediction is possible to have a sufficient effect of reducing the dose when combining the two neuromuscular blocking agents through monitoring neuromuscular relaxation during surgery.

METHODS: Each group were intubating dose group (Group I, n=27) combined Effective Dose (ED)95 rocuronium and ED95 cisatracurium, small amount reducing group (Group S, n=27) reduced 10% of each ED95 and large amount reducing group (Group L, n=27) reduced 20% of each ED95. Before patients arrived in the operating room, rocuronium and cisatracurium were prepared by a nurse who was not involved in this study. Each study drug was administrated to the patient and timer was started with TOF-Watch® monitoring. Train-of-four (TOF) of the ulnar nerve was used as setting of 2 Hz per 12 sec. The investigators checked time to TOF ratio=0 (Onset), time to 1st TOF ratio>25% (Duration 25%) and TOF 25-75% (recovery index) under total i.v. anesthesia (TIVA). One way ANOVA was used for statistical analysis (α=0.05, β=0.2).

DETAILED DESCRIPTION:
Introduction:

Rocuronium and cisatracurium are representative neuromuscular blocking agents used widely because the former have features of fast onset of peak effect and short duration of muscle relaxation relatively while the latter have comparatively long duration relaxation time and break down by Hofmann elimination and ester hydrolysis. A combination of the two have a synergic effect may be also used with either the priming method for rapid sequence intubation. It would contribute both to determine the effective combination rate clinically and to predict the pharmacokinetic characteristics that determine how much the synergistic effect of this combination. The investigators studied whether the prediction is possible to have a sufficient effect of reducing the dose when combining the two muscle relaxants through monitoring muscle relaxation during surgery.

Materials and methods:

This study was conducted to 81 patients scheduled for elective mastoidectomy and tympanoplasty after obtaining written informed consent. All patients included the American Society of Anesthesiologists (ASA) physical status I-II, aged 20-60, BMI 20-30 kg/m2. The exclusion criteria were as follows: a history of allergy to the study drugs, neuromuscular disease, pregnancy or breast-feeding, preoperative medication of antipsychotics or neuroleptics known to interact with non-depolarizing neuromuscular blocking agents (NMBAs), serum creatinine level>1.2 mg/dL, liver transaminase>40 U/L. Anthropometric variables such as height, weight were measured in ward before surgery. BMI calculated as total body weight divided by the squared height. Ideal body weight (IBW) was calculated by the formula of Devine {50 kg + 2.3 × (height [inch]-60) for man and 45.5 kg + 2.3 × (height [inch]-60) for woman} and used to administrate NMBAs of initial dose. Lean body weight (LBW) was calculated by the formula of James {LBW (men) = (1.10 × Weight(kg)) - 128 × ( Weight2 / (100 × Height(m))2), (women) = (1.07 × Weight(kg)) - 148 × ( Weight2 / (100 × Height(m))2)}. Additive dose of NMBAs was administrated by LBW. Patients were randomly assigned to each group by opening of sealed allocation envelope. Each group were intubating dose group (Group I, n=27) combined ED95 rocuronium and ED95 cisatracurium, small amount reducing group (Group S, n=27) reduced 10% of each ED95 and large amount reducing group (Group L, n=27) reduced 20% of each ED95.

Monitoring and Medication:

In the operating room, monitoring was accomplished to patients with a noninvasive blood pressure, pulse oximetry, electrocardiography, thermometer, Bispectral Index (BIS VISTA Monitoring System; Aspect Medical Systems Inc, Norwood, MA, USA), and T1/T4 ratio used TOF-Watch® (Organon, Teknica B.V., Boxtel, the Netherlands). Every 5 min, measured things are recorded.

Premedications with midazolam 2 mg and glycopyrrolate 0.2 mg were administrated to patients intramuscularly 1 h before surgery. Before patients arrived in the operating room, rocuronium and cisatracurium were prepared by a nurse who was not involved in this study. The syringe containing each study drug was conveyed to the performer of this study as the status of shielding the scale. The syringes of rocuronium and cisatracurium used each other syringe. Anesthesia was induced with propofol 1.5-2.5 mg/kg, remifentanil 0.4-0.6 mcg/kg, afterward maintained with target controlled infusion (TCI) of propofol 5-10 mg/kg/hr and remifentanil 0.05-2 mcg/kg/min. The infusion pump (Orchestra Module DPS, Fresenius-Vial, Brezins, France) was operated with Minto's and Marshall's pharmacokinetic model for effect site TCI of remifentanil and propofol.

The opposite arm against operation side was used for neuromuscular monitoring and attached to armboard of TOF-Watch®. Each study drug was administrated to the patient and timer was started with T1/T4 ratio monitoring. The surface electrodes of ulnar nerve placed at the wrist and Train-of-four (TOF) stimulation was used as setting of supramaximal square wave impulses with 200μs duration, 2 Hz per 12sec. The investigators checked times to TOF ratio=0 (Onset), 1st TOF ratio>25% (Duration 25%) and TOF 25-75% (Recovery Index), recovery time of 90% (TOF 25-90%) under total i.v. anesthesia (TIVA). Also the investigators checked the rate of additional rescue dose administrated with 10% of initial NMBAs dose, operation time from incision to surgical wound dressing, anesthesia time from entering to going out the operation room. Body temperature was maintained above 35°C using warm air blanket. The arterial pressure cuff was placed on the opposite arm against TOF monitoring.

Adverse Events and Management:

In all patients, anesthesia level was assessed based on a BIS score of 40-60. Moderate hypertension (>120% of baseline) or hypotension (<80% of baseline) was treated by increasing or decreasing rate of propofol infusion with fluid supplement. Severe hemodynamic change (systolic pressure < 90 mmHg or > 200 mmHg) was controlled by intravenous (IV) administration of phenylephrine 50 mcg or nicardipine 250 mcg repeatedly until being hemodynamic stable status. Unexpectedly, when hiccup or self-contained respiration was showed, additional rescue dose of NMBAs was administrated to the patient even though T1/T4 ratio was lower than 25%.

Statistical Analysis:

All data are expressed as means ± standard deviations (SDs), numbers (percentages), or medians (upper and lower quartiles), as appropriate. Data between the groups were compared using the χ2 test, Fisher exact test, independent t test, or the Mann-Whitney U test, as appropriate. To assess data normality, the Kolmogorov-Smirnov test was performed on the data set. According to a preliminary study, 24 patients would be required in each group with a power of 0.9 and a type I error of 0.05. Factoring in a drop-out rate of 10%, the investigators calculated that 27 patients would be required for each group. All statistical analyses were performed with the SPSS 18.0 (SPSS Inc., Chicago, IL, USA) program. A P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* the American Society of Anesthesiologists (ASA) physical status I-II
* BMI 20-30 kg/m2
* Patients scheduled for mastoidectomy and tympanoplasty.

Exclusion Criteria:

* a history of allergy to the study drugs,
* neuromuscular disease,
* pregnancy
* breast-feeding,
* preoperative medication of antipsychotics or neuroleptics known to interact with NMBAs
* serum creatinine level>1.2 mg/dL,
* liver transaminase>40 U/L.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young Gwan Cheon, Study Director — Institutional Review Board of Wonju Severance Christian Hospital

REFERENCES:
- [Background] Naguib M, Samarkandi AH, Ammar A, Elfaqih SR, Al-Zahrani S, Turkistani A. Comparative clinical pharmacology of rocuronium, cisatracurium, and their combination. Anesthesiology. 1998 Nov;89(5):1116-24. doi: 10.1097/00000542-199811000-00011. PMID 9821999
- [Background] Donati F, Plaud B. Rocuronium-cisatracurium combinations. Anesthesiology. 1999 Aug;91(2):587-8. doi: 10.1097/00000542-199908000-00054. No abstract available. PMID 10443637
- [Background] Miller DR, Wherrett C, Hull K, Watson J, Legault S. Cumulation characteristics of cisatracurium and rocuronium during continuous infusion. Can J Anaesth. 2000 Oct;47(10):943-9. doi: 10.1007/BF03024863. PMID 11032267
- [Background] Cammu G, de Baerdemaeker L, den Blauwen N, de Mey JC, Struys M, Mortier E. Postoperative residual curarization with cisatracurium and rocuronium infusions. Eur J Anaesthesiol. 2002 Feb;19(2):129-34. doi: 10.1017/s0265021502000236. PMID 11999596
- [Background] Hans P, Welter P, Dewandre PY, Brichant JF, Bonhomme V. Recovery from neuromuscular block after an intubation dose of cisatracurium and rocuronium in lumbar disc surgery. Acta Anaesthesiol Belg. 2004;55(2):129-33. PMID 15264506
- [Background] Mak PH, Irwin MG. The effect of cisatracurium and rocuronium on cisatracurium precurarization and the priming principle. J Clin Anesth. 2004 Mar;16(2):83-7. doi: 10.1016/j.jclinane.2003.05.004. PMID 15110367
- [Background] Kopman AF, Zank LM, Ng J, Neuman GG. Antagonism of cisatracurium and rocuronium block at a tactile train-of-four count of 2: should quantitative assessment of neuromuscular function be mandatory? Anesth Analg. 2004 Jan;98(1):102-106. doi: 10.1213/01.ANE.0000094985.19305.E9. PMID 14693596
- [Background] de Morais BS, de Castro CH, Teixeira VC, Pinto AS. Residual neuromuscular block after rocuronium or cisatracurium. Rev Bras Anestesiol. 2005 Dec;55(6):622-30. doi: 10.1590/s0034-70942005000600005. English, Portuguese. PMID 19468536
- [Background] Kopman AF, Kopman DJ, Ng J, Zank LM. Antagonism of profound cisatracurium and rocuronium block: the role of objective assessment of neuromuscular function. J Clin Anesth. 2005 Feb;17(1):30-5. doi: 10.1016/j.jclinane.2004.03.009. PMID 15721727
- [Background] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- [Background] Adamus M, Gabrhelik T, Marek O. Influence of gender on the course of neuromuscular block following a single bolus dose of cisatracurium or rocuronium. Eur J Anaesthesiol. 2008 Jul;25(7):589-95. doi: 10.1017/S026502150800402X. Epub 2008 Apr 11. PMID 18405411
- [Background] Lin SP, Chang KY, Chen YJ, Lin SM, Chang WK, Chan KH, Ting CK. Priming with rocuronium to accelerate the onset time of cisatracurium during intubation. J Chin Med Assoc. 2009 Jan;72(1):15-9. doi: 10.1016/S1726-4901(09)70014-0. PMID 19181592
- [Background] Amin AM, Mohammad MY, Ibrahim MF. Comparative study of neuromuscular blocking and hemodynamic effects of rocuronium and cisatracurium under sevoflurane or total intravenous anesthesia. Middle East J Anaesthesiol. 2009 Feb;20(1):39-51. PMID 19266825
- [Background] Fassbender P, Geldner G, Blobner M, Hofmockel R, Rex C, Gautam S, Malhotra A, Eikermann M. Clinical predictors of duration of action of cisatracurium and rocuronium administered long-term. Am J Crit Care. 2009 Sep;18(5):439-45. doi: 10.4037/ajcc2009883. PMID 19723864
- [Background] Lee H, Jeong S, Choi C, Jeong H, Lee S, Jeong S. Anesthesiologist's satisfaction using between cisatracurium and rocuronium for the intubation in the anesthesia induced by remifentanil and propofol. Korean J Anesthesiol. 2013 Jan;64(1):34-9. doi: 10.4097/kjae.2013.64.1.34. Epub 2013 Jan 21. PMID 23372884
- [Result] Leykin Y, Pellis T, Lucca M, Lomangino G, Marzano B, Gullo A. The pharmacodynamic effects of rocuronium when dosed according to real body weight or ideal body weight in morbidly obese patients. Anesth Analg. 2004 Oct;99(4):1086-1089. doi: 10.1213/01.ANE.0000120081.99080.C2. PMID 15385355
- [Result] Breslin DS, Jiao K, Habib AS, Schultz J, Gan TJ. Pharmacodynamic interactions between cisatracurium and rocuronium. Anesth Analg. 2004 Jan;98(1):107-110. doi: 10.1213/01.ANE.0000093387.15263.48. PMID 14693597
- [Result] Leykin Y, Pellis T, Lucca M, Gullo A. Intubation conditions following rocuronium: influence of induction agent and priming. Anaesth Intensive Care. 2005 Aug;33(4):462-8. doi: 10.1177/0310057X0503300407. PMID 16119487
- [Result] Kim KS, Chun YS, Chon SU, Suh JK. Neuromuscular interaction between cisatracurium and mivacurium, atracurium, vecuronium or rocuronium administered in combination. Anaesthesia. 1998 Sep;53(9):872-8. doi: 10.1046/j.1365-2044.1998.00492.x. PMID 9849281
- [Result] Liu M, Dilger JP. Synergy between pairs of competitive antagonists at adult human muscle acetylcholine receptors. Anesth Analg. 2008 Aug;107(2):525-33. doi: 10.1213/ane.0b013e31817b4469. PMID 18633030
- [Result] Zeidan A, Nahle N, Maaliki H, Baraka A. Cisatracurium or rocuronium versus rocuronium-cisatracurium combination. Middle East J Anaesthesiol. 2006 Jun;18(5):879-86. PMID 17094524
- [Result] Lighthall GK, Jamieson MA, Katolik J, Brock-Utne JG. A comparison of the onset and clinical duration of high doses of cisatracurium and rocuronium. J Clin Anesth. 1999 May;11(3):220-5. doi: 10.1016/s0952-8180(99)00030-6. PMID 10434218
- [Derived] Park WY, Choi JC, Yun HJ, Jeon YG, Park G, Choi JB. Optimal dose of combined rocuronium and cisatracurium during minor surgery: A randomized trial. Medicine (Baltimore). 2018 Mar;97(10):e9779. doi: 10.1097/MD.0000000000009779. PMID 29517695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Started | 27 | 27 | 27
Completed | 27 | 27 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L | Total
Number analyzed (Participants) | 27 | 27 | 27 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (10.7) | 50.3 (8.0) | 49.3 (9.4) | 49.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 20 | 56
  Male | 9 | 9 | 7 | 25
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 27 | 27 | 27 | 81

OUTCOME MEASURES:

1. Primary Outcome: Onset of Neuromuscular Blocking Agents(NMBAs)
Description: Time from administration of initial NMBAs to Train-of-four (TOF) ratio=0, assessed up to 15 minutes during general anesthesia.
Time Frame: Intraoperative, an average of 5 minutes
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Second | 212.8 (56.0) | 230.1 (60.6) | 399.3 (147.8)

2. Primary Outcome: Duration 25% of Neuromuscular Blocking Agents(NMBAs)
Description: Time from administration of initial NMBAs to Train-of-four (TOF) ratio >25%, assessed up to 2 hours during general anesthesia.
Time Frame: Intraoperative, an average of 1 hours
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Minute | 51.3 (8.4) | 47.9 (10.7) | 39.4 (6.8)

3. Primary Outcome: Recovery Index of Neuromuscular Blocking Agents(NMBAs)
Description: Time from TOF ratio 25% to 75%, assessed up to 1 hour during general anesthesia.
Time Frame: Intraoperative, an average of 20 minutes
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Minute | 15.9 (3.8) | 16.2 (4.8) | 14.1 (3.4)

4. Secondary Outcome: Operation Time
Description: Time from skin incision to wound dressing assessed up to 8 hours.
Time Frame: Intraoperative, an average of 3 hours.
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Minute | 151.8 (27.2) | 147.0 (31.4) | 145.9 (27.6)

5. Secondary Outcome: Anesthetic Time
Description: Time from induction to recovery of anesthesia, asessed up to 3 hours.
Time Frame: Intraoperative, an average 4 hours.
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Minute | 163.0 (26.8) | 159.9 (30.6) | 161.4 (25.9)

6. Secondary Outcome: Additional Rescue Doses Per Hour Ratio.
Description: Additional Rescue Doses Per Hour Ratio is the number per hour of addition of rescue dose administrated with 10% of initial NMBAs dose. The formula is {(Addition number + 1 / Anesthetic time) x 60}.
Time Frame: Intraoperative, an average of 3 hours.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
ratio | 1.43455 (0.49108) | 1.21014 (0.43501) | 0.82128 (0.26596)

7. Other Pre Specified Outcome: Non Invasive Blood Pressure,
Description: Before induction of anesthesia, non invasive blood pressure was measured for baseline.
  And after injection of NMBAs, non invasive blood pressure was measured at 10 min.
Time Frame: Before and after induction of anesthesia, an average 10 min.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
mmHg
  Systolic pressure | 128.3 (17.7) | 128.3 (20.7) | 128.4 (19.1)
  Diastolic pressure | 75.6 (9.7) | 76.7 (9.2) | 74.8 (9.0)

8. Other Pre Specified Outcome: Peripheral Oxygen Saturation
Description: Before induction of anesthesia, peripheral oxygen saturation was measured for baseline.
  And after injection of NMBAs, peripheral oxygen saturation was measured at 10 min.
Time Frame: Before and after induction of anesthesia, an average 10 min.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Percentage | 100 (0.0) | 99.9 (0.2) | 100 (0.0)

9. Other Pre Specified Outcome: Body Temperature
Description: Before induction of anesthesia, body temperature was measured for baseline by oral temperature probe.
  And after injection of NMBAs, non invasive blood pressure was measured at 10 min by esophageal temperature probe.
Time Frame: Before and after induction of anesthesia, an average 10 min.
Measure: Mean (Standard Deviation); unit: Celcius degree
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
Celcius degree | 36.3 (0.3) | 36.3 (0.2) | 36.3 (0.2)

10. Other Pre Specified Outcome: Bispectral Index
Description: The BIS monitor provides a single dimensionless number, which ranges from 0 (equivalent to EEG silence) to 100. A BIS value between 40 and 60 indicates an appropriate level for general anesthesia, as recommended by the manufacturer.
  Before induction of anesthesia, bispectral index was measured for baseline. And after injection of NMBAs, bispectral index was measured at 10 min.
Time Frame: Before and after induction of anesthesia, an average 10 min.
Measure: Mean (Standard Deviation); unit: BIS score
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
Number analyzed (Participants) | 27 | 27 | 27
BIS score | 46.0 (8.2) | 46.1 (7.5) | 44.3 (9.4)

ADVERSE EVENTS:
Time Frame: Adverse events are divided to intraoperative adverse events and postoperative adverse events. Intraoperative adverse events are collected until end of anesthesia. And postoperative adverse events are collected from end of anesthesia to 1 month (until next visiting outpatient clinic after discharge).
Groups:
- Intubating Dose, Group I: combined ED95 rocuronium and ED95 cisatracurium
  ED95, dose causing on average 95% suppression of neuromuscular response.
  The duration of intubation did not differ between groups. Group I and S were intubation Grade 0 (Excellent) intubation.
- 10% Reduction of Combination of Esmeron® and Nimbex®, Group S: This arm reduced 10% of combined ED95 rocuronium and ED95 cisatracurium
  10% reduction of combination of Esmeron® and Nimbex®: Patients were randomly assigned to each group by opening of sealed allocation envelope. After collection of data, allocation number was matched with each group. The participants matched at Group S were administered with NMBAs reduced 10% of each ED95. Before patients arrived in the operating room, rocuronium and cisatracurium were prepared by a nurse who was not involved in this study. Each drug dosage was determined by allocation number. The syringe containing each study drug was conveyed to the performer of this study as the status of shielding the scale. The syringes of rocuronium and cisatracurium used each other syringe.
  The duration of intubation did not differ between groups. Group I and S were intubation Grade 0 (Excellent) intubation
- 20% Reduction of Combination of Esmeron® and Nimbex®, Group L: This arm reduced 20% of combined ED95 rocuronium and ED95 cisatracurium
  20% reduction of combination of Esmeron® and Nimbex®: The participants matched at Group L were administered with NMBAs reduced 20% of each ED95.
  Group L included 1 patient with Grade 1 (Good) intubation and 2 patients with Grade 2 (Poor) intubation. The patients with Grade 2 intubation coughed during intubation and 1 of these patients produced small arm movements during coughing.
Arm/Group | Intubating Dose, Group I | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3.7% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intubating Dose, Group I (N=27) | 10% Reduction of Combination of Esmeron® and Nimbex®, Group S (N=27) | 20% Reduction of Combination of Esmeron® and Nimbex®, Group L (N=27)
Coughing (Investigations) | 0 (0) | 0 (0) | 2 (2) — Patient had weak coughing reflex during intubation.
Agitation (Investigations) | 0 (0) | 0 (0) | 1 (1) — Patient had weak involuntary movement of hand during intubation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No